CLINICAL TRIAL: NCT00472667
Title: Impact of Procalcitonin to Reduce Antibiotics Use in ICU Adults Patients
Brief Title: PROcalcitonin Reduce Antibiotic Treatments in Acute-Ill Patients (PRORATA)
Acronym: PRORATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Aurelie GUIMFACK, Department Clinical Research of Developpement
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: P060204; AOR06019
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2007-05

CONDITIONS: Bacterial Infections
Keywords: Bacterial infections; Procalcitonin; Intensive care unit; Antibiotic therapy; Suspicion of bacterial infection or proven
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Procalcitonin guided strategy
  Interventions: Procedure: Procalcitonin guided strategy

INTERVENTIONS:
Procedure: Procalcitonin guided strategy — Procalcitonin guided strategy

SUMMARY:
The study is a prospective, randomized, controlled intervention trial conducted in 9 centers, comparing a conventional strategy versus a PCT-guided strategy to start or to discontinue antibiotics, in patients with suspected community or hospital- acquired infection.

DETAILED DESCRIPTION:
Clinical and laboratory signs are neither specific nor sensitive for diagnosis of sepsis in critically-ill patients. Because delaying antimicrobial therapy may be deleterious, broad-spectrum antibiotics are widely used in ICU -patients, even when they are not needed. In addition, only few well-designed studies concerning the duration of antibiotic treatment have been so far published. Consequently, many patients received antibiotics during the ICU stay. Many studies have shown that exposure to antibiotics, the so called "selection pressure" is an independent risk factor for acquisition of resistance in individual patients. Therefore, reducing antibiotic use is probably necessary to control antibiotic resistance. Many clinical studies have shown that procalcitonin (PCT) is able to distinguish the inflammatory response to infection from other types of inflammation and to distinguish bacterial from viral infections. Recent studies have shown that PCT guidance substantially and safely reduced antibiotic overuse in patients with lower respiratory tract infections. We aimed to evaluate the role of PCT in reducing the use of antibiotics in ICU adult patients. The study is a prospective, randomized, controlled intervention trial conducted in 9 centers, comparing a conventional strategy versus a PCT-guided strategy to start or to discontinue antibiotics, in patients with suspected community or hospital- acquired infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised in the ICU
* Bacterial infection suspected
* At ICU admission the patient do not receive antibiotics or receive antibiotics for less than 24hours and an interval between admission and inclusion < 12 hours
* During ICU stay, provided that the interval between the start of suspected infection and inclusion is < 12hours
* Written inform consent from the patient or relatives. The consent may be obtained after the enrollment if the patient is not able to give consent and if there is no relatives

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Patient expected to remain hospitalised in the ICU for less than 3 days
* Neutropenia
* Infection or presumed infection requiring prolonged antibiotic therapy (endocarditis,osteo-articular infection, mediastinitis, deep abscess, tuberculosis, pneumocystis pneumonia, toxoplasmosis).
* Simplified Acute Physiology Score II at ICU admission (calculated during the first 12h)
* Attending physician declining to use full life support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Exposition to antibiotics, defined by antibiotic-free days | assessed 28 days after inclusion
Mortality | at Day 28 and Day 60

SECONDARY OUTCOMES:
Consumption of antibiotics expressed as the Defined Daily Dose/1000 ICU-days | between D1 and D28
The length of ICU and hospital stay | during the stay at the hospital
The evolution of SOFA score parameters | between D1 and D28
The number of mechanical ventilation-free days | at D28
The acquisition cost of antibiotics | between D1 and D28
The percentage of emerging multiresistant bacteria between D1 and D28, as assessed by microbiologic examination of all clinical samples. | between D1 and D28
The percentages of relapses of infection | between D1 and D28

CONTACTS AND LOCATIONS:
Overall Officials: Lila BOUADMA, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Chu Bichat Claude Bernard, Paris, France

REFERENCES:
- [Derived] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417